CLINICAL TRIAL: NCT00806728
Title: Phase I Study of MEDI-507 in the Treatment of Adult Patients With at Least Grade II Steroid-Resistant Acute Graft-Versus-Host Disease
Brief Title: Study of MEDI-507 in With Steroid-Resistant Acute Graft-Versus-Host Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: J. Bruce McClain, M.D., Medimmune Inc.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MI-CP042
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Last update posted 2008-12-11 (Estimated); Status verified 2008-12

CONDITIONS: Cancer; Graft-Versus-Host Disease
MeSH Terms: conditions — Neoplasms; Graft vs Host Disease | interventions — siplizumab

ARMS (2):
- 1 (Experimental): MEDI-507
  Interventions: Drug: MEDI-507
- 2 (Experimental): MEDI-507
  Interventions: Drug: MEDI-507

INTERVENTIONS:
Drug: MEDI-507 — 0.12 mg/kg of MEDI-507 given every third day for 4 doses followed by doses of normal saline on Days 16, 23, 30, and 37.
  Arms: 1
Drug: MEDI-507 — 0.12 mg/kg of MEDI-507 given every third day for 4 doses followed by doses of MEDI-507 on Days 16, 23, 30, and 37.
  Arms: 2

SUMMARY:
A clinical trial to assess safety and two regimens of (MEDI-507) a drug given to stem cell and bone marrow recipients who have a mid-grade acute Graft-versus-Host Disease.

DETAILED DESCRIPTION:
To assess the safety of two regimens of MEDI-507 administered to stem cell and bone marrow allograft recipients who have at least grade II acute GVHD and who have not achieved a satisfactory response to at least three days of corticosteroid therapy (2 mg/kg/day of methylprednisolone or its equivalent).

ELIGIBILITY:
Inclusion Criteria:

* Allogeneic bone marrow or hematopoietic stem cell graft recipients
* Acute GVHD of at least grade II severity
* Failure of GVHD to improve on at least 2 mg/kg/day of methylprednisolone or prednisone for at least three days or recurrence of acute GVHD as corticosteroids are tapered from initial treatment of the initial episode of GVHD
* Evidence of engraftment (ANC over 1000 cells/mm3)
* Histologic evidence of GVHD from biopsy performed during the current episode
* Received GVHD prophylaxis of methotrexate, tacrolimus or cyclosporine
* Age at least 18 years
* Body weight under 130 kg
* Both males and females are eligible but females of childbearing potential will use an accepted method of avoiding pregnancy for at least 60 days after the end of treatment (which includes oral or implanted contraceptives, IUD, female condom, diaphragm with spermicide, cervical cap, abstinence, use of a condom by the sexual partner or a sterile sexual partner)

Exclusion Criteria:

* Previous receipt of MEDI-507
* Clinical or histologic manifestation of chronic GVHD
* Previous treatment with any anti-T-cell antibodies such as OKT®3 or daclizumab (Zenapax®)
* Receipt of antithymocyte globulin (ATGAM® or other ATG) since the day of transplant
* More than one allogeneic bone marrow or hematopoietic stem cell allograft
* Moribund and unlikely (in the opinion of the investigator) to survive 15 days
* Use of other investigational agents within 30 days (this does not include the use of licensed agents for indications not listed in the package insert)
* Any of the following clinical settings or diagnoses:

Ø documented or presumed significant active infection Ø pregnancy or nursing mother Ø evidence of infection with HIV-1, hepatitis B or C virus Ø hemodialysis or chronic peritoneal dialysis Ø use of a ventilator

* Histologically confirmed veno-occlusive disease of the liver
* Ascites on physical examination (this does not include small amounts of ascitic fluid detected only on ultrasound)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 1998-05; Primary Completion 1998-11 (Actual); Study Completion 1998-12 (Actual)

PRIMARY OUTCOMES:
Safety was assessed by the direct observation of patients, medical history, and clinical laboratory evaluation to determine the incidence of patients experiencing AEs. | Day 0-60

SECONDARY OUTCOMES:
Pharmacokinetics, Lymphocyte Phenotype and CD2 Receptor Occupancy Pharmacodynamics | Study Days 12 and 44

CONTACTS AND LOCATIONS:
Overall Officials: J. Bruce McClain, M.D., Study Director — MedImmune LLC
Locations (10):
- United States (10):
  - City of Hope National Medical Center, Duarte, California
  - University of Colorado Health Sciences Center, Denver, Colorado
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Washington University Medical Center, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Hospital-University of Oklahoma, Oklahoma City, Oklahoma
  - Western Pennsylvania Hospital - Western Pennsylvania Cancer Center, Pittsburgh, Pennsylvania
  - Baylor University Medical Center, Dallas, Texas
  - M.D. Anderson Cancer Center, Houston, Texas
  - South Texas Cancer Institute at Methodist Hospital, San Antonio, Texas